CLINICAL TRIAL: NCT02131987
Title: Radiological Riskfactors for Dislocation of Hip Hemiarthroplasty Through a Posterolateral Approach as Treatment for Femoral Neck Fracture
Brief Title: Radiological Riskfactors for Dislocation of Hip Hemiarthroplasty
Acronym: RRDHHR
Status: Completed | Type: Observational
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SMASN; SM
Record Dates: First submitted 2014-04-28; First posted 2014-05-06 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Dislocation; Femoral Neck Fracture
Keywords: Dislocation; Hemiarthroplasty; Femoral neck fracture; Femoral offset; Leg length difference; Wiberg angle
MeSH Terms: conditions — Joint Dislocations; Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dislocation: Patients operated with hip hemiarthroplasty for a femoral neck fracture with a postoperative dislocation of the prosthesis
- Non-dislocated: Patents without dislocation of a hemiarthroplasty for a femoral neck fracture

SUMMARY:
Between January 1 2006 and December 31 2013, at our department 324 patients underwent hemiarthroplasty (HA) for displaced femoral-neck fracture with a bipolar prosthesis (Variokopf, Link®, Germany) by the use of the posteriolateral approach. Patients with pathological fractures and HA performed with direct lateral approach were excluded. A retrospective cohort study were conducted. Patients with prosthetic dislocation formed one group and patients without dislocation formed the control group.

As standard, post surgery radiographs (anteroposterior and lateral) were taken. After these were performed patient started weight bearing as soon as possible. Clinical data regarding patient demographics, details of the surgical procedure and the medical comorbidities were collected by the use of patient and operative records. Radiological analysis with position evaluation was performed using the post surgery radiographs by measuring Wiberg angle, inequality of leg length and femoral offset of the prostheses and compared with non-operated hip joint using the post surgery x-ray images.

Our hypothesis were that patients with single- or recurrent dislocations had shortened postoperative leg length, decreased femoral offsed and a Wiberg angle less than 25 degrees.

ELIGIBILITY:
Inclusion Criteria:

* Femoral neck fracture
* Treated with Hemiarthroplasty
* Through a posterolateral approach

Exclusion Criteria:

* Direct lateral approach

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between January 1 2006 and December 31 2013, at our department 324 patients underwent hemiarthroplasty (HA) for displaced femoral-neck fracture with a bipolar prosthesis (Variokopf, Link®, Germany) by the use of the posteriolateral approach. Patients with pathological fractures and HA performed with anterolateral approach were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2006-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Femoral offset | 6 months up to 7 years
  The femoral offset is measured on the postoperative X-ray. The result are compared between the groups of dislocated and non-dislocated patients.
Leg length difference | 6 months to 7 years
  Leg length difference is measured on the postoperative X-ray. The result are compared between the groups of dislocated and non-dislocated patients.
Wiberg angle | 6 months to 7 years
  Wiberg angle is measured on the postoperative X-ray. The result are compared between the groups of dislocated and non-dislocated patients.

SECONDARY OUTCOMES:
1 year mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: Arkan S Sayed-Noor, MD,PhD,FRCS, Principal Investigator — Orthopaedic department, Sundsvalls sjukhus, Landstinget Västernorrland
Locations (1):
- Orthopaedic department, Sundsvall hospital, Sundsvall, Västernorrland County, Sweden

REFERENCES:
- [Background] Madanat R, Makinen TJ, Ovaska MT, Soiva M, Vahlberg T, Haapala J. Dislocation of hip hemiarthroplasty following posterolateral surgical approach: a nested case-control study. Int Orthop. 2012 May;36(5):935-40. doi: 10.1007/s00264-011-1353-0. Epub 2011 Sep 20. PMID 21931967
- [Background] Ninh CC, Sethi A, Hatahet M, Les C, Morandi M, Vaidya R. Hip dislocation after modular unipolar hemiarthroplasty. J Arthroplasty. 2009 Aug;24(5):768-74. doi: 10.1016/j.arth.2008.02.019. Epub 2008 Jun 13. PMID 18555648
- [Background] Enocson A, Pettersson H, Ponzer S, Tornkvist H, Dalen N, Tidermark J. Quality of life after dislocation of hip arthroplasty: a prospective cohort study on 319 patients with femoral neck fractures with a one-year follow-up. Qual Life Res. 2009 Nov;18(9):1177-84. doi: 10.1007/s11136-009-9531-x. Epub 2009 Aug 28. PMID 19714486
- [Result] Mukka S, Lindqvist J, Peyda S, Broden C, Mahmood S, Hassany H, Sayed-Noor A. Dislocation of bipolar hip hemiarthroplasty through a postero-lateral approach for femoral neck fractures: A cohort study. Int Orthop. 2015 Jul;39(7):1277-82. doi: 10.1007/s00264-014-2642-1. Epub 2015 Jan 6. PMID 25557759